CLINICAL TRIAL: NCT02891304
Title: A Prospective Multi-center Randomized Controlled Trial Evaluating Endoscopy Competence Among Gastroenterology Trainees in the Era of the Next Accreditation System.
Brief Title: Trial Evaluating Endoscopy Competence Among Gastroenterology Trainees in the Era of the Next Accreditation System.
Acronym: EnCompAS
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: University of California, Los Angeles (Other); University of California, Irvine (Other); Drexel University College of Medicine (Other); University of South Alabama (Other); The University of Texas Health Science Center at San Antonio (Other); Northwestern University (Other); University Hospitals Cleveland Medical Center (Other); Advocate Lutheran General Hospital (Other); Washington University School of Medicine (Other); Emory University (Other); Rush University (Other); Ochsner Health System (Other); St. John Providence Health System (Other); University of Wisconsin, Madison (Other); State University of New York - Downstate Medical Center (Other); University of North Carolina (Other); University of Miami (Other); New York Medical College (Other)
Responsible Party: Sponsor
Other Study IDs: 16-0782
Record Dates: First submitted 2016-08-29; First posted 2016-09-07 (Estimated); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Competency in General Endoscopic Surgical Procedures
Keywords: esophagogastroduodenoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Quarterly Feedback: In addition to each center's traditional endoscopic feedback for trainees, centers/trainees will receive objective feedback every 3-months on trainee overall performance including learning curves on ACE tool performance, performance relative to de-identified anonymous peers on each of the individual skills (e.g. fine tip control), and the global assessment for technical and cognitive skill achievement. For those skills which are not advanced/superior - trainees will additionally receive links to online didactic videos which teach these skills.
  Interventions: Other: Quarterly Feedback
- Annual Feedback: In addition to each center's traditional endoscopic feedback for trainees, centers/trainees will receive learning curves at the end of each training year. Learning curves, relative to de-identified anonymous peers will be provided to program directors annually (June).

INTERVENTIONS:
Other: Quarterly Feedback — Learning curves received quarterly vs. annually
  Groups: Quarterly Feedback

SUMMARY:
Hypothesis: ACE (The Assessment in Competency in Endoscopy Tool) tool for colonoscopy and EGD (Esophagogastroduodenoscopy) allows for reliable standardized learning curves, competency benchmarks, and creation of a centralized database that compares trainee performance amongst peers. Trainees receiving quarterly learning curves achieve competence in endoscopic procedures at a faster rate (ie less procedures) compared to trainees receiving usual feedback on endoscopic performance as established by their respective GI (gastrointestinal) fellowship program.

Aims: To compare the number of procedures necessary to achieve competence in EGD and colonoscopy between trainees receiving learning curve performance feedback every three months in addition to standard feedback versus trainees receiving annual learning curve performance feedback in addition to standard feedback for these endoscopic procedures. To demonstrate the feasibility of development and adoption of a centralized database that would allow program directors and general GI trainees to generate performance reports in relation to national peers to provide real-time targeted performance feedback during training and evaluate trainee and GI fellowship program directors predictors of competence.

DETAILED DESCRIPTION:
There has been an increasing emphasis on standardizing competency assessment and demonstrating readiness for independent practice as medical training transitions from an apprenticeship model to competency based medical education (CBME). The Accreditation Council for Graduate Medical Education (ACGME) replaced their long-standing reporting system in 2014 with the Next Accreditation System (NAS). For Gastroenterology (GI) fellowship programs (GIFPs), this includes assessing and documenting competence in basic endoscopic procedures [esophagogastroduodenoscopy (EGD)] in a continuous fashion. For colonoscopy, the prior minimum threshold of 140 procedures after which competence can be assessed was based on surrogates of competence such as cecal intubation rate, with limited assessment of technical and cognitive skills required to perform high-quality endoscopic examination. Recent data has demonstrated wide variability in trainee learning curves, hence emphasis needs to be shifted away from the volume of procedures performed to independent performance of well-defined metrics. Tools with comprehensive assessment of motor and cognitive abilities have been developed. The American Society for Gastrointestinal Endoscopy (ASGE) endorsed the assessment of competence in endoscopy tool (ACE) designed to help GIFPs facilitate implementation of the NAS requirements. While the ACE tool for EGD has yet to be validated, Sedlack and colleagues recently validated the ACE tool in colonoscopy. Multicenter prospective data are needed to help guide development of CBME that define learning curves in colonoscopy and EGD and generate a centralized database which will allow programs to provide individualized feedback and follow trainee performance longitudinally throughout training.

ELIGIBILITY:
Inclusion Criteria:

* Attendings and trainees in GI Fellowship Program

Exclusion Criteria:

* N/A

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Attendings and trainees in GI Fellowship Program
Sampling Method: Non-Probability Sample
Enrollment: 157 (Actual)
Dates: Start 2016-07; Primary Completion 2018-06-15 (Actual); Study Completion 2018-06-15 (Actual)

PRIMARY OUTCOMES:
ACE Tool Validation | 3 years
  Primary Aim: Using the ACE tool with a comprehensive electronic data collection and reporting system, the primary aim of this study is to compare the number of procedures necessary to achieve competence in EGD and colonoscopy between trainees receiving learning curve performance feedback every three months in addition to standard feedback as provided by supervising attendings at a given institution versus trainees receiving annual learning curve performance feedback in addition to standard feedback for these endoscopic procedures as provided by supervising attendings at a given institution.

SECONDARY OUTCOMES:
Development of Centralized Performance Database | 3 years
  To demonstrate the feasibility of development and adoption of a centralized database that would allow program directors and general GI trainees to generate performance reports in relation to national peers to provide real-time targeted performance feedback during training and evaluate trainee and GIFP predictors of competence.

CONTACTS AND LOCATIONS:
Overall Officials: Sachin Wani, MD, Principal Investigator — University of Colorado, Denver

REFERENCES:
- [Derived] Han S, Obuch JC, Keswani RN, Hall M, Patel SG, Menard-Katcher P, Simon V, Ezekwe E, Aagaard E, Ahmad A, Alghamdi S, Austin K, Brimhall B, Broy C, Carlin L, Cooley M, Di Palma JA, Duloy AM, Early DS, Ellert S, Gaumnitz EA, Goyal J, Kathpalia P, Day L, El-Nachef N, Kerman D, Lee RH, Lunsford T, Mittal M, Morigeau K, Pietrak S, Piper M, Shah AS, Shapiro AB, Shergill A, Sonnier W, Sorrell C, Vignesh S, Wani S. Effect of individualized feedback on learning curves in EGD and colonoscopy: a cluster randomized controlled trial. Gastrointest Endosc. 2020 Apr;91(4):882-893.e4. doi: 10.1016/j.gie.2019.10.032. Epub 2019 Nov 9. PMID 31715173